CLINICAL TRIAL: NCT06676670
Title: Huazhong University of Science and Technology
Brief Title: Discussion on the Mechanism of Acupuncture on Patients with Paroxysmal Migraine Without Aura : a Randomized Controlled Clinical Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bo Huang (Other)
Responsible Party: Sponsor-Investigator, Bo Huang, Teaching secretary, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021MWOATJ01
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-02

CONDITIONS: Migraine, Dysmenorrhea
MeSH Terms: conditions — Migraine Disorders; Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- real acupuncture group (Experimental): 1. The patient immediately received acupuncture treatment and imaging scan on the scanning bed (acupuncture and imaging scan at the same time). Acupuncture left Hegu point to promote qi. Axial T2WI imaging for 48 seconds, fMR-BOLD imaging for 8 minutes and 11 seconds, and ASL imaging for 6 minutes and 03 seconds were simultaneously collected during acupuncture. The scanning time of each sequence was divided into 4 time periods, each time period was 1 time, each scanning sequence was 4 times, each time was 10 seconds, and the duration of acupuncture was 15 minutes and 02 seconds.
  2. After acupuncture withdrawal, axial T2WI imaging was repeated for 48 seconds, fMRI-Bold imaging for 8 minutes and 11 seconds, and ASL imaging for 6 minutes and 03 seconds.
  Interventions: Other: real acupuncture
- sham acupuncture group (Sham Comparator): Control group (false acupuncture group)
  1. Axial imaging of DWI was performed before the patient underwent pseudoacupuncture (12 minutes 08 seconds).
  2. The patient immediately underwent a sham acupuncture and imaging scan on the scanning bed (the sham acupuncture and imaging scan were performed simultaneously). Pseudoacupuncture left Hegu point. DWI axial imaging (12 minutes 08 seconds) was collected synchronously during the fake acupuncture. The scanning time during the fake acupuncture was divided into 4 time periods, with 1 needle in each time period, 4 needles in each time period, each time for 10 seconds, and the duration of the fake acupuncture was 12 minutes 08 seconds.
  3. Axial DWI imaging was repeated (12 minutes and 08 seconds) after acupuncture withdrawal.
  Interventions: Other: sham acupuncture
- healthy controls (No Intervention)

INTERVENTIONS:
Other: real acupuncture — Real Acupuncture Group Main acupoints: Hegu (bilateral), Taichong (bilateral), Taiyang (unilateral), shuogu (unilateral), Fengchi (unilateral); Positioning: refer to the 2006 national standard of the people's Republic of China (gb/t 12346-2006) acupoint names and positioning Operation method: supine position, skin routine disinfection. The special model of acupuncture and moxibustion (0.30mm × 30mm), fix the gasket on the acupoint skin with seam free tape, and then acupuncture. After acupuncture, each acupoint will be lifted, inserted and twisted three times in small amplitude; The needle will be kept for 30 minutes. During this period, the technique of small amplitude uniform lifting, inserting and twisting (3 times) will be performed every 10 minutes. A total of four times of needling will be performed.
  Arms: real acupuncture group
Other: sham acupuncture — Sham acupuncture group Acupoint selection: select eight stimulation points at the neck and shoulder. Stimulation point 1: the midpoint of the line between the shoulder well and the giant bone (both sides); Stimulation point 2: 5 inches (both sides) of the inferior paraspinal process of the seventh thoracic vertebra; Stimulus point 3: the inferior paraspinal process of the eighth thoracic vertebra will be opened 5 inches (bilateral); Stimulus point 4: 5 inches (both sides) of the infraspinous process of the ninth thoracic vertebra.
  Positioning: refer to the 2006 national standard of the people's Republic of China (gb/t 12346-2006) acupoint names and positioning to avoid acupoints.
  Operation method: supine position, skin routine disinfection. Streitberger acupuncture (0. 300×30mm). Fix the gasket on the acupoint skin with seam free tape,and then acupuncture. After acupuncture, each acupoint will be lifted, inserted and twisted three times in small amplitude; The needle will be kept fo
  Arms: sham acupuncture group

SUMMARY:
Background: Migraine is common but poorly managed with drugs. Acupuncture, a non-pharmacological approach, has shown promise, yet its mechanisms remain unclear. This study aims to assess the efficacy and specificity of acupuncture for acute paroxysmal migraine without aura.

Methods: A randomized, single-blind, sham-controlled trial will recruit 60 patients from Tongji Hospital, China. Patients will receive 20 sessions of Deqi or sham acupuncture over 4 weeks and be followed for 8 weeks. Treatments will occur twice within 4 hours of headache onset. Primary outcome is complete headache remission within 120 minutes after two treatments without analgesics. Secondary outcomes include headache intensity reduction, remission rates, and adverse events. Blind assessment will be conducted after at least one session. Data will be analyzed using full and per-protocol sets.

Ethics: Approved by the Clinical Trial Ethics Committee (approval no: TJ-IRB20220573). Written consent will be obtained. Results will be published in a peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* 1\They met the diagnostic criteria of migraine without aura and had a history ofmore than 1 year; 2\Age 18-65 years old;

  * 18.5kg/m2 ≤ BMI ≤ 30.0kg / m2,right-handed; ④ The average frequency of migraine attacks in recent 6 months was ≥ 2-8 times per month; The average number of migraine attacks per month in recent 6 months was less than 15 days; The neurological examination was negative, and the CT or MRI of the head was normal; There was no experience of acupuncture or migraine prevention and treatment in recent 3 months; Able to complete the baseline migraine diary; Agree to sign the informed consent form.

Exclusion Criteria:

* Other types of primary headache or secondary headache; It is complicated with serious primary diseases such as cardiovascular,cerebrovascular, liver, kidney, gastrointestinal, blood, nervous system, etc; Complicated with severe mental illness; In the past 12 weeks, migraine drugs were taken orally or headache treatment methods such as acupuncture and physiotherapy were received; Lactation, pregnant women and planned pregnant women; Participate in another clinical trial at the same time; Illiterate, unable to read comprehension scale; Poor compliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2026-02-19 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of people with complete remission of migraine | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China